CLINICAL TRIAL: NCT00512915
Title: Atriale Vorhofsonde 1699 Mit Sehr Kurzem Bipolabstand Zur Vermeidung Von Far Field Sensing
Brief Title: Avoid FFS - Use of the Atrial Pacemaker Lead 1699 With Very Short Tip Ring Spacing to Avoid Far Field Sensing
Acronym: Avoid FFS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Jörg Scheiner, St. Jude Medical GmbH
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: B84
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Atrial Fibrillation; Bradycardia
Keywords: Farfield Sensing; Pacing lead; Postventricular atrial blanking; Bradycardia
MeSH Terms: conditions — Atrial Fibrillation; Bradycardia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1699T (Optisense) (Active Comparator): Implantation of the Optisense Lead 1699T, programming of the shortest possible postventricular atrial blanking period (PVAB)
  Interventions: Device: pacemaker implantation
- Standard lead (Active Comparator): Implantation of a standard bipolar atrial pacing lead. Optimization of the postventricular atrial blanking period (PVAB) after implantation.
  Interventions: Device: pacemaker implantation

INTERVENTIONS:
Device: pacemaker implantation — St. Jude Medical Dual Chamber Pacemaker model Identity (ADx) DR, Victory DR, or newer
  Other Names: Active Arm: 1699T Tendril Optisense lead; Standard lead: 1688T Tendril SDX, 1788T Tendril ST, 1888T Tendril ST OPTIM

SUMMARY:
The purpose of this study is to evaluate the possibility to program the shortest possible Post Ventricular Atrial Blanking Period (PVAB) and high sensitivity without getting inappropriate Mode Switch due to Far Field R-Wave sensing when using the new Tendril 1699T lead. Comparison with Tendril 1688T or 1388T with optimized Post Ventricular Atrial Blanking (PVAB).

DETAILED DESCRIPTION:
Far-field R-wave sensing (FFS) in the atrial channel of dual chamber pacemakers is a relevant source for inappropriate Mode Switch from the DDD mode to the DDI or VDI mode. Inappropriate loss of atrioventricular synchrony due to false positive Mode Switch is hemodynamically disadvantageous, may induce atrial tachyarrhythmias, can lead to pacemaker syndrome, and impairs the reliability of pacemaker Holter data. The aim of the study is to determine whether the use of a new atrial screw in lead with ultra short tip-ring distance of 1.1 mm (Study Group) eliminates the need for individual adjustment of the postventricular atrial blanking period (PVAB) based on an additional test in the Control Group with standard leads.

ELIGIBILITY:
Inclusion Criteria:

* Indication for dual chamber pacing
* Implantation of an Identity (ADX) DR or Victory or later pacemaker (St. Jude Medical)
* Bipolar atrial pacing electrode
* Age >= 18 years

Exclusion Criteria:

* Persistent / permanent Atrial Arrhythmia
* Pacemaker Revision
* Pregnancy
* Participation in another Study involving active implantable medical devices
* Unable to complete follow up
* Missing patient informed consent
* Cardiac surgery or myocardial infarction within the last 4 weeks
* Planned cardiac surgery within 3 months after enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2006-12; Primary Completion 2008-05 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Incidence of inappropriate mode switch (documented by stored EGM's) using the atrial lead Tendril 1699T with short post ventricular atrial blanking period (PVAB) compared to standard atrial lead (Tentril 1388 or 1688) with optimised PVAB | 1 and 3 months post implantation

SECONDARY OUTCOMES:
Incidence of inappropriate mode switch in respect to lead position and ventricular stimulation frequency | 1 and 3 months post implantation
Atrial Flutter in stored EGM's | 1 and 3 months post implantation
2:1 lock in of Atrial Flutter | 1 and 3 months post implantation

CONTACTS AND LOCATIONS:
Overall Officials: Christof Kolb, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (10):
- Germany (10):
  - Klinikum Coburg, Coburg
  - Klinik Fränkische Schweiz, Ebermannstadt
  - Kreisklinik Ebersberg, Ebersberg
  - Krankenhaus Waltershausen-Friedrichroda, Friedrichroda
  - Universitäres Herzzentrum Hamburg, Hamburg
  - Klinikum Memmingen, Memmingen
  - Deutsches Herzzentrum Muenchen, Munich
  - Kardiologische Praxis Dres. med. Bödigheimer / Mühling / Prof. Dr. med. Silber, München
  - Kreiskrankenhaus Ottweiler, Ottweiler
  - Universitätsklinikum Ulm, Ulm

REFERENCES:
- [Derived] Kolb C, Nolker G, Lennerz C, Jetter H, Semmler V, Purner K, Gutleben KJ, Reents T, Lang K, Lotze U; AVOID-FFS Investigators. Use of an atrial lead with very short tip-to-ring spacing avoids oversensing of far-field R-wave. PLoS One. 2012;7(6):e38277. doi: 10.1371/journal.pone.0038277. Epub 2012 Jun 22. PMID 22745661